CLINICAL TRIAL: NCT02243930
Title: Cap-assisted Sigmoidoscopy - Reduction in Pain, Reduction in Investigation Time and Increased Rate of Success, When Examined by the Less-experienced Endoscopist. A Prospective Randomized Clinical Trial
Brief Title: Cap-assisted Sigmoidoscopy - Influence on Pain, Duration and Rate of Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, magnus Ploug, MD, Junior Doctor, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: KOESURG-41580; 41580 (Other: The regional committee of health research ethics)
Record Dates: First submitted 2014-09-12; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Pain
Keywords: Sigmoidoscopy with or without cap; Pain during sigmoidoscopy; Sigmoidoscopy and time
MeSH Terms: conditions — Pain | interventions — Contraceptive Devices, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cap (Experimental): Sigmoidoscopy with cap
  Interventions: Device: Disposable distal attachment
- No cap (No Intervention): Sigmoidoscopy without cap

INTERVENTIONS:
Device: Disposable distal attachment
  Other Names: "cap"; Model No. D-201-14304 - Olympus; Dimentions: Ø15,0mm
  Arms: Cap

SUMMARY:
The purpose of this study is to investigate the attachment of a transparent hood ("cap") on the sigmoidoscope. The investigators hypothesis is that this will reduce pain, reduce investigation time, and increases the success rate of the sigmoidoscopy. The study focus on the less-experienced endoscopist.

DETAILED DESCRIPTION:
The investigators randomize study subject to sigmoidoscopy +/- the attachment of the cap.

Using a 100mm VAS scale the investigators record pain when the sigmoidoscopy reaches its intubation end-point (60cm from anus). The investigators also register the time spent to this point and the rate of examinations not achieving this endpoint.

ELIGIBILITY:
Inclusion Criteria:

* planned to undergo sigmoidoscopy
* informed consent

Exclusion Criteria:

* use of iv medication for pain and/or anxiety immediately before the endoscopy
* lack of indication for a full sigmoidoscopy (eg just need to investigate the rectum)
* lack or improper administration of standard bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
VAS recording of pain | During endoscopy. The subject is randomized immediately prior to the endoscopy. The outcome measures are all measured during examination.
  the registration is performed when the endoscopist has advanced the scope to the 60 cm mark.

SECONDARY OUTCOMES:
Time | During endoscopy. The subject is randomized immediately prior to the endoscopy. The outcome measures are all measured during examination.
  Recording of the time it takes from the introduction of the endoscopy through anus until it reaches 60 cm intubation mark.

OTHER OUTCOMES:
rate of success | During endoscopy. The subject is randomized immediately prior to the endoscopy. The outcome measures are all measured during examination.
  recording the rate of examinations that reached the intubation endpoint at 60cm from anus

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Ploug, MD, Principal Investigator — Koege Hospital, Surgical Department
Locations (1):
- Surgical department, endoscopy unit, Koege Hospital, Denmark, Koege, Region Sjælland, Denmark

REFERENCES:
- [Derived] Ploug M, Poulsen JK, Jensen HQ, Achiam M. The use of a transparent cap in sigmoidoscopy-A randomized controlled clinical trial on pain, time and success rate. Indian J Gastroenterol. 2017 Jul;36(4):318-322. doi: 10.1007/s12664-017-0776-y. Epub 2017 Aug 1. PMID 28762140